CLINICAL TRIAL: NCT05001880
Title: Phase 2 Randomized Trial of Neoadjuvant or Palliative Chemotherapy With or Without Immunotherapy for Peritoneal Mesothelioma
Brief Title: Chemotherapy With or Without Immunotherapy for Peritoneal Mesothelioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-08573; NCI-2021-08573 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A092001 (Other: Alliance for Clinical Trials in Oncology); A092001 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2021-08-11; First posted 2021-08-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Peritoneal Malignant Mesothelioma
MeSH Terms: interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Carboplatin; Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy; Pemetrexed; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (carboplatin, pemetrexed, bevacizumab, atezolizumab) (Experimental): Patients receive atezolizumab IV over 30-60 minutes, bevacizumab IV over 30-90 minutes, carboplatin IV over 30 minutes, and pemetrexed IV over 10 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 4-8 weeks, patients then undergo cytoreductive surgery and HIPEC. Patients not eligible for surgery may receive atezolizumab IV over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 1 of each maintenance therapy cycle. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan, PET scan, and collection of blood and tissue samples throughout the study.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Cytoreductive Surgery; Drug: Hyperthermic Intraperitoneal Chemotherapy; Drug: Pemetrexed; Procedure: Positron Emission Tomography
- Arm II (carboplatin, pemetrexed, bevacizumab) (Active Comparator): Patients receive bevacizumab IV over 30-90 minutes, carboplatin IV over 30 minutes, and pemetrexed IV over 10 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 4-8 weeks, patients then undergo cytoreductive surgery and HIPEC. Patients not eligible for surgery may receive bevacizumab IV over 30-90 minutes with or without atezolizumab IV over 30-60 minutes on day 1 of each maintenance therapy cycle at the discretion of the investigator. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan, PET scan, and collection of blood and tissue samples throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Cytoreductive Surgery; Drug: Hyperthermic Intraperitoneal Chemotherapy; Drug: Pemetrexed; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm I (carboplatin, pemetrexed, bevacizumab, atezolizumab)
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Cytoreductive Surgery — Undergo surgery
  Other Names: Cytoreduction
Drug: Hyperthermic Intraperitoneal Chemotherapy — Undergo HIPEC
  Other Names: HIPEC
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial compares the usual treatment alone (carboplatin, pemetrexed, and bevacizumab) to using immunotherapy (atezolizumab) plus the usual treatment in treating patients with peritoneal mesothelioma. The usual treatment consists of surgery or chemotherapy. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of cancer cells. Pemetrexed is in a class of medications called antifolate antineoplastic agents. It works by stopping cells from using folic acid to make deoxyribonucleic acid and may kill cancer cells. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving atezolizumab with usual treatment may work better than usual treatment alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether frontline treatment with carboplatin, pemetrexed, bevacizumab and atezolizumab results in a superior best response rate than carboplatin, pemetrexed and bevacizumab in patients with peritoneal mesothelioma as determined by Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OBJECTIVES:

I. To determine the safety, major pathologic response rates, and completeness of cytoreduction of patients treated with neoadjuvant carboplatin, pemetrexed, bevacizumab and atezolizumab or carboplatin, pemetrexed and bevacizumab.

II. To determine the safety of patients treated with palliative carboplatin, pemetrexed, bevacizumab and atezolizumab or carboplatin, pemetrexed and bevacizumab.

III. To determine whether frontline treatment with carboplatin, pemetrexed, bevacizumab and atezolizumab results in a superior metabolic response rate than carboplatin, pemetrexed and bevacizumab as determined by Positron Emission Tomography (PET) Response Criteria in Solid Tumors.

IV. Explore the value that analysis of secondary computed tomography (CT) findings and quantitative fludeoxyglucose F-18 (FDG)-PET imaging adds to prognostic information and response assessment in this disease.

V. Determine the number of patients who were deemed to have unresectable disease who are able to undergo surgery following treatment with carboplatin, pemetrexed, bevacizumab and atezolizumab or carboplatin, pemetrexed and bevacizumab due to dramatic response.

VI. To compare the progression-free survival and overall survival between arms. VII. Results of the primary analysis will be examined for consistency, while taking into account the stratification factors and/or covariates of baseline quality of life (QOL) and fatigue.

EXPLORATORY OBJECTIVE:

I. To determine whether blood-based biomarkers including our recently described cell-free chromosomal junctions, soluble mesothelin-related peptides and megakaryocyte potentiating factor correlate with clinical outcomes data (i.e. overall survival [OS], progression-free survival [PFS], recurrence, response, etc.).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive atezolizumab intravenously (IV) over 30-60 minutes, bevacizumab IV over 30-90 minutes, carboplatin IV over 30 minutes, and pemetrexed IV over 10 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 4-8 weeks, patients then undergo cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (HIPEC). Patients not eligible for surgery may receive atezolizumab IV over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 1 of each maintenance therapy cycle. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive bevacizumab IV over 30-90 minutes, carboplatin IV over 30 minutes, and pemetrexed IV over 10 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 4-8 weeks, patients then undergo cytoreductive surgery and HIPEC. Patients not eligible for surgery may receive bevacizumab IV over 30-90 minutes with or without atezolizumab IV over 30-60 minutes on day 1 of each maintenance therapy cycle at the discretion of the investigator. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients also undergo CT scan, PET scan, and collection of blood and tissue samples throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Physicians should consider whether any of the following may render the patient inappropriate for this protocol:

  * Psychiatric illness which would prevent the patient from giving informed consent
  * Medical conditions such as uncontrolled infection, uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient

    * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
    * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
    * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
  * Patients with a "currently active" second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for >= 3 years
* In addition:

  * Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives or double barrier method (diaphragm plus condom)

    * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Histologically or cytologically confirmed malignant peritoneal mesothelioma for which there has been no prior treatment. Given the indolent nature of well-differentiated papillary mesothelioma and multicystic mesothelioma, patients with these variants are not eligible for participation
* Must have measurable disease per RECIST version (v) 1.1
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 28 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Leukocytes >= 2,500/mm^3
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine clearance >= 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) =< 3.0 x upper limit of normal (ULN)
* Urine protein/creatinine (UPC) ratio < 1, or urine protein: =< 1+
* No prior systemic therapy for peritoneal mesothelioma is allowed. No concurrent radiotherapy is allowed
* No active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

  * Rash must cover < 10% of body surface area
  * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
  * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* No history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* No prior allogeneic stem cell or solid organ transplantation
* Central nervous system (CNS) metastases must have been treated with local therapy (surgery, radiation, ablation) with systemic steroids tapered to a physiologic dose (10 mg or prednisone equivalent or less)
* Patients who have received live attenuated vaccines within 30 days of the first dose of trial treatment are eligible at the discretion of the investigator. All seasonal influenza vaccines and vaccines intended to prevent SARS-CoV-2 and coronavirus disease 2019 (COVID-19) are allowed
* No history of inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* No history of hypertensive crisis or hypertensive encephalopathy
* No clinically significant cardiovascular disease, such as cerebrovascular accidents within 12 months prior to randomization, myocardial infarction within 12 months prior to randomization, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with study treatment
* No significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to randomization
* No history of grade >= 4 venous thromboembolism
* No history or evidence upon physical or neurological examination of central nervous system disease (e.g. seizures) unrelated to cancer unless adequately treated with standard medical therapy
* No history of grade >= 2 hemoptysis (defined as >= 2.5 mL of bright red blood per episode) within 1 month prior to screening
* No history or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
* No major surgical procedure or significant traumatic injury within 28 days prior to initiation of study treatment (diagnostic laparoscopy is allowed as part of diagnosing peritoneal mesothelioma)
* No core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to initiation of study treatment
* Placement of a vascular access device should be at least 2 days prior to initiation of study treatment
* No active infection requiring IV antibiotics at the time of initiation of study treatment
* No history of abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess, or active GI bleeding within 6 months prior to randomization
* No serious, non-healing wound, active ulcer, or untreated bone fracture
* No other malignancy within 5 years prior to randomization, except for localized cancer in situ, such as basal or squamous cell skin cancer
* Patients with a creatinine clearance between 45 and 79 mL/min should not use ibuprofen or other nonsteroidal anti-inflammatory drug (NSAIDs) for 2 days before, the day of, and 2 days following pemetrexed administration
* No treatment with immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) may be eligible for the study
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 4 years after study activation
  Will be compared between arms.

SECONDARY OUTCOMES:
Major pathologic response rate | Up to 3 years
  The proportion of patients with a pathologic response will be calculated and compared between arms and 95% confidence intervals reported. The chi-square test will be used to compare the rates between arms.
Completeness of cytoreduction | Up to 3 years
  Will be estimated.
Conversion rate to surgical resection among those not deemed to be surgical candidates | Up to 3 years
  Will estimate the conversion rate to surgical resection among those not deemed to be surgical candidates prior to treatment and provide the 95% confidence interval as well.
Progression-free survival (PFS) | From study entry to the first of either disease progression or death from any cause, where disease progression will be determined based on Response Evaluation Criteria in Solid Tumors 1.1 criteria, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.
Overall survival | From study entry to death from any cause, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.
Incidence of adverse events | Up to 3 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events version 5.0. The frequency and percentage of grade 3+ adverse events will be compared between the 2 treatment arms. Comparisons between arms will be made by using either the Chi-square or Fisher's Exact test.

OTHER OUTCOMES:
Soluble mesothelin-related peptides and megakaryocyte potentiating factor | Up to 3 years
  Will be correlated with clinical endpoints including confirmed response, overall survival, PFS, recurrence, and adverse events. Statistical and graphical techniques will be used to explore the relationships between the translational and clinical data. For time-to-event endpoints, will use Cox proportional hazards models, and for confirmed response will use Logistic regression models. In addition, will use the Chi-square or Fisher's exact tests to test the association between categorical marker data and confirmed response/adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Mansfield, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (39):
- United States (39):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Alliance for Clinical Trials in Oncology, Boston, Massachusetts
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Steadman JA, Grotz TE. Principles of Surgical Management of Peritoneal Mesothelioma. J Natl Compr Canc Netw. 2023 Sep;21(9):981-986. doi: 10.6004/jnccn.2023.7055. PMID 37673112